CLINICAL TRIAL: NCT07122232
Title: Comparative Analysis of Thrombocytopenia in Plasmodium Vivax and Plasmodium Falciparum Malaria: A Prospective Cross-Sectional Study From a Tertiary Care Hospital in Peshawar, Pakistan
Brief Title: Comparative Study of Thrombocytopenia in Plasmodium Vivax and Falciparum Malaria
Status: Completed | Type: Observational
Sponsor: Rafiullah Hotak (Other)
Collaborators: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Sponsor-Investigator, Rafiullah Hotak, Student, Nangarhar University
Organization: Nangarhar University (Other)
Other Study IDs: Ref: No. 617/LRH/MTI
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Malaria; Plasmodium Vivax Infection; Plasmodium Falciparum Infection; Thrombocytopenia
Keywords: Thrombocytopenia; Plasmodium falciparum; Malaria complications; Platelet count dynamics
MeSH Terms: conditions — Malaria; Thrombocytopenia; Malaria, Falciparum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Plasmodium vivax Group: Adult patients (≥18 years) with microscopically confirmed Plasmodium vivax malaria. Platelet counts and clinical data were collected at admission, day 3, and day 7 to assess the frequency and severity of thrombocytopenia.
- Plasmodium falciparum Group: Adult patients (≥18 years) with microscopically confirmed Plasmodium falciparum malaria. Platelet counts and clinical data were collected at admission, day 3, and day 7 to assess the frequency and severity of thrombocytopenia.

SUMMARY:
This study aimed to compare platelet count patterns in patients infected with either Plasmodium vivax or Plasmodium falciparum, the two most common malaria species in Pakistan. Thrombocytopenia (low platelet count) is a common complication of malaria and can help in identifying disease severity. We conducted this research at a tertiary care hospital in Peshawar, Pakistan, from April to September 2023. A total of 171 adult patients with confirmed malaria infections were enrolled. We measured their platelet counts at admission, day 3, and day 7, and analyzed the severity and progression of thrombocytopenia. The study found that while P. vivax was more common, P. falciparum was more likely to cause severe thrombocytopenia. Understanding these differences helps healthcare providers identify high-risk patients earlier and manage malaria more effectively. The study was approved by the institutional review board of Lady Reading Hospital, Peshawar.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Microscopically confirmed infection with Plasmodium vivax or Plasmodium falciparum
* Provided written informed consen

Exclusion Criteria:

* Mixed-species malaria infection
* Known hematologic disorders
* Chronic liver disease
* Recent blood transfusion
* Use of anticoagulant medication
* Incomplete parasitemia data or lost to follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18 and above) presenting to a tertiary care hospital in Peshawar, Pakistan, with confirmed malaria infection. Participants were included based on microscopic confirmation of either Plasmodium vivax or Plasmodium falciparum infection and evaluated for platelet trends and clinical outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with thrombocytopenia | 0 days
  The percentage of patients with platelet counts <50×10³/µL at admission, compared between the P. vivax and P. falciparum groups.

SECONDARY OUTCOMES:
Platelet count recovery over time | Day 0 to Day 7
  Change in mean platelet count at admission, day 3, and day 7, for each group.

OTHER OUTCOMES:
Frequency of malaria-related complications | Within 7 days of admission
  Number of patients developing clinical complications (e.g., acute kidney injury, neurological involvement, anemia, jaundice), stratified by malaria species.

CONTACTS AND LOCATIONS:
Overall Officials: Rafiullah Hotak, MBBS, Principal Investigator — Nangarhar University faculty of medicine
Locations (1):
- Lady Reading Hospital, Medical Teaching Institution, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No